CLINICAL TRIAL: NCT00693693
Title: Adherence to Topical Hydrocortisone 17-butyrate 0.1% (Locoid®) Using Different Vehicles in Adults With Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00000702
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Results first posted 2017-03-17 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — hydrocortisone-17-butyrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cream- (Active Comparator): topical hydrocortisone 17-butyrate 0.1% Cream preparation applied twice daily to all lesions of atopic dermatitis
  Interventions: Drug: hydrocortisone 17-butyrate 0.1% Cream preparation
- Ointment (Active Comparator): topical hydrocortisone 17-butyrate 0.1% Ointment preparation applied twice daily to all lesions of atopic dermatitis
  Interventions: Drug: hydrocortisone 17-butyrate 0.1% Ointment preparation
- Lipocream (Active Comparator): topical hydrocortisone 17-butyrate 0.1% Lipocream preparation applied twice daily to all lesions of atopic dermatitis
  Interventions: Drug: hydrocortisone 17-butyrate 0.1% Lipocream preparation

INTERVENTIONS:
Drug: hydrocortisone 17-butyrate 0.1% Cream preparation — Apply medication twice a day to affected areas of atopic dermatitis
  Other Names: Locoid
  Arms: Cream-
Drug: hydrocortisone 17-butyrate 0.1% Ointment preparation — Apply medication twice a day to affected areas of atopic dermatitis
  Other Names: locoid
  Arms: Ointment
Drug: hydrocortisone 17-butyrate 0.1% Lipocream preparation — Apply medication twice a day to affected areas of atopic dermatitis
  Other Names: locoid
  Arms: Lipocream

SUMMARY:
The purpose of this research study is to better understand adherence to Locoid when people use it to treat atopic dermatitis.

DETAILED DESCRIPTION:
An investigator-blinded prospective study of subjects with mild to moderate atopic dermatitis (>5% Body Surface area and 2 or 3 on the Investigator Global Assessment (IGA) scale). The drug will be used within FDA-approved labeling. Subjects will be randomized to each of the following topical hydrocortisone 17-butyrate 0.1% preparations- ointment, cream or lipocream- in the manufacturer's original tube fitted with a Medication Event Monitoring System (MEMS) cap. This cap records dates and times the assembly is opened and this data can be downloaded and tabulated with the associated software.

The study will consist of a 2-week Treatment Phase (visits at Baseline and Week 2). Subjects will be instructed to apply the medication twice daily (morning and evening) for 2 weeks to all of their AD lesions.

Adherence will be measured by MEMs cap.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age.
* Subjects must have diagnosis of mild to moderate atopic dermatitis using IGA criteria. (2 or 3 on severity scale)
* Subjects must have >5% TBSA and <30% to be enrolled.
* Women of child bearing potential will be allowed to participate in the study, and these subjects will be required to use at least one form of birth control.

Exclusion Criteria:

* Known allergy or sensitivity to topical Locoid® cream, ointment or lipocream in the subject.
* Inability to complete all study-related visits.
* Introduction of any other prescription medication, topical or systemic, for atopic dermatitis while participating in the study.
* Requiring >130 gm of cream in a 2 week period.
* Having facial or groin involvement of their disease.
* Pregnant women and women who are breast feeding are to be excluded. Women of child bearing potential will be allowed to participate in the study, and these subjects will be required to use at least one form of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-11; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Feldman, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Dermatology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from IRB approved advertising and the Dermatology Clinic.
Groups:
- Ointment: topical hydrocortisone 17-butyrate 0.1% preparation ointment
- Lipocream: topical hydrocortisone 17-butyrate 0.1% preparation lipocream
- Cream: topical hydrocortisone 17-butyrate 0.1% preparation cream
Period: Overall Study
Arm/Group | Ointment | Lipocream | Cream
Started | 7 | 9 | 9
Completed | 6 | 8 | 7
Not Completed | 1 | 1 | 2
Not completed — Lost to Follow-up | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Cream: topical hydrocortisone 17-butyrate 0.1% cream applied twice daily
- Ointment: topical hydrocortisone 17-butyrate 0.1% ointment applied twice daily
- Lipocream: topical hydrocortisone 17-butyrate 0.1% Lipocream applied twice daily
- Total: Total of all reporting groups
Arm/Group | Cream | Ointment | Lipocream | Total
Number analyzed (Participants) | 9 | 7 | 9 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 7 | 9 | 25
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 5 | 14
  Male | 4 | 3 | 4 | 11
Region of Enrollment [Number; unit: participants]
  United States | 9 | 7 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Locoid
Description: Adherence measured by MEMS cap as the % of days that the two total prescribed doses were applied
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: percentage of days
Groups:
- Cream: topical hydrocortisone 17-butyrate 0.1% cream applied twice daily to all areas of atopic dermatitis
- Ointment: topical hydrocortisone 17-butyrate 0.1% ointment applied twice daily to all areas of atopic dermatitis
- Lipocream: topical hydrocortisone 17-butyrate 0.1% Lipocream applied twice daily to all areas of atopic dermatitis
Arm/Group | Cream | Ointment | Lipocream
Number analyzed (Participants) | 6 | 7 | 8
percentage of days | .55 (.07) | .60 (.07) | .50 (.07)

ADVERSE EVENTS:
Groups:
- Topical Hydrocortisone 17-butyrate 0.1% Cream: topical hydrocortisone 17-butyrate 0.1% cream applied twice daily
- Topical Hydrocortisone 17-butyrate 0.1% Ointment: topical hydrocortisone 17-butyrate 0.1% ointment applied twice daily
- Topical Hydrocortisone 17-butyrate 0.1% Lipocream: topical hydrocortisone 17-butyrate 0.1% lipocream applied twice daily
Arm/Group | Topical Hydrocortisone 17-butyrate 0.1% Cream | Topical Hydrocortisone 17-butyrate 0.1% Ointment | Topical Hydrocortisone 17-butyrate 0.1% Lipocream
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No